CLINICAL TRIAL: NCT02344654
Title: Fluorescence Cholangiography Versus X-ray Cholangiography During Laparoscopic Cholecystectomy for Complicated Gallstone Disease
Brief Title: Fluorescence Cholangiography During Cholecystectomy - a RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Lars Lang Lehrskov, MD, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2015-HVH-LLS-01
Record Dates: First submitted 2015-01-09; First posted 2015-01-26 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Cholecystitis; Gallstones
Keywords: Fluorescence; Cholangiography; Indocyanine Green; Cholecystectomy, Laparoscopic
MeSH Terms: conditions — Cholecystitis; Gallstones | interventions — Indocyanine Green; Diatrizoate Meglumine; X-Rays

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fluorescence cholangiography (Experimental): After induction of anaesthesia 2.5-7.5 mg of indocyanine green (0.05 mg/kg) is injected intravenously. The operation field is routinely inspected in the fluorescence imaging mode before dissection of Calot´s triangle. During dissection, the fluorescence imaging mode is used when needed, before division of any tubular structure and after division of the cystic duct and artery.
  Interventions: Drug: Indocyanine green; Device: Near-infrared illumination
- X-ray cholangiography (Active Comparator): The cholangiography is performed after dissection of the cystic duct by cannulation of the cystic duct with a catheter using either a Kumar- or Olsen grasper. A mobile X-ray C-arm system is used, and the monochrome X-ray image is shown on a separate screen. After satisfactory identification of the extra-hepatic biliary ducts, the intraoperative cholangiography is discontinued and the gallbladder is removed in a standardized manner.
  Interventions: Drug: Urografin; Radiation: X-ray

INTERVENTIONS:
Drug: Indocyanine green
  Arms: Fluorescence cholangiography
Device: Near-infrared illumination — To see the fluorescence from indocyanine green
  Arms: Fluorescence cholangiography
Drug: Urografin
  Arms: X-ray cholangiography
Radiation: X-ray
  Arms: X-ray cholangiography

SUMMARY:
The primary objective is to compare the success rates of intraoperative fluorescent cholangiography using indocyanine green versus conventional X-ray cholangiography for the identification of bile duct anatomy during laparoscopic cholecystectomy for complicated gallstone disease in a randomized design with 120 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for planned laparoscopic cholecystectomy by one surgeon
* Complicated gallstone disease

Exclusion Criteria:

* Open cholecystectomy
* Allergy towards iodine, urografin or indocyanine green
* Liver or renal insufficiency
* Thyrotoxicosis
* Pregnancy or lactation
* Legally incompetent for any reason
* Withdrawal of inclusion consent at any time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2018-08-27 (Actual)

PRIMARY OUTCOMES:
Visualization of the cystic duct - common hepatic duct - common bile duct junction | Intraoperative

SECONDARY OUTCOMES:
Time spend for intraoperative fluorescent cholangiography/conventional X-ray cholangiography | Intraoperative
Surgeon satisfaction score (Measured on a 5 point VAS scale) | Intraoperative
  Measured on a 5 point VAS scale
Per-/postoperative adverse events as a measure of safety and tolerability | Intraoperative
Total cost of operation incl fluorescent/conventional X-ray cholangiography | Admission to discharge from hospital (0-30 days)

CONTACTS AND LOCATIONS:
Overall Officials: Lars ML Lehrskov-Schmidt, MD, Principal Investigator — Hvidovre University Hospital

REFERENCES:
- [Result] Lehrskov LL, Westen M, Larsen SS, Jensen AB, Kristensen BB, Bisgaard T. Fluorescence or X-ray cholangiography in elective laparoscopic cholecystectomy: a randomized clinical trial. Br J Surg. 2020 May;107(6):655-661. doi: 10.1002/bjs.11510. Epub 2020 Feb 14. PMID 32057103
- [Derived] Lehrskov LL, Larsen SS, Kristensen BB, Bisgaard T. Fluorescence versus X-ray cholangiography during laparoscopic cholecystectomy: protocol for a randomised trial. Dan Med J. 2016 Aug;63(8):A5261. PMID 27477798